CLINICAL TRIAL: NCT04018846
Title: The Future of the Revascularization Using a Bioprotec Graft
Brief Title: The Future of Revascularization Using a Bioprotec Graft
Acronym: REVATEC
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0518
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Revascularization; Graft; Vein; Artery; Limb; Amputation
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Revascularization using a BIOPROTEC Graft — It is about a routine care study not changing the usual follow-up of patients: postoperative visits after a Doppler ultrasonography made by a vascular Doctor in 1 month, 6 months, 12 months, 18 months and 2 years.
  Other Names: BIOPROTEC Vascular Graft

SUMMARY:
The main purpose of this study is the rate assessment of rescued limbs, one year after a BIOPROTEC vascular graft.

DETAILED DESCRIPTION:
The BIOPROTEC grafts are controverted: they are useful in some cases, but they are known as frequently broken or thrombosed. However they are always posed in a complicated situations, in a fragile patients who have ever had many of revascularizations or in an infectious state (which is supportive of the pseudoaneurysm and thrombosis) Despite the frequent use of this graft in France, the results have never been published.

ELIGIBILITY:
Inclusion Criteria:

* ≥ Eighteen years old.
* Critical ischemia (Phase 4-6 of Rutherford): no saphenous equipment for the vascular reconstruction; at least one leg axis permeable.

Exclusion Criteria:

* Pregnant woman.
* Patient with an acute ischemia.
* Patient with an exceeded ischemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Grafted patient with a vascular BIOPROTEC graft in case of a Peripheral artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
The Limb rescue rate one year after a BIOPROTEC graft | Two years
  Usual follow-up of patients: postoperative visits after a Doppler ultrasonography made by a vascular doctor in 1 month, 6 months, 12 months, 18 months and 2 years

SECONDARY OUTCOMES:
The revascularization permeability rate | Two years
  Usual follow-up of patients: postoperative visits after a Doppler ultrasonography made by a vascular doctor in 1 month, 6 months, 12 months, 18 months and 2 years
The amputation rate | Two years
  Usual follow-up of patients: postoperative visits after a Doppler ultrasonography made by a vascular doctor in 1 month, 6 months, 12 months, 18 months and 2 years
Infection resistance rate | Two years
  Usual follow-up of patients: postoperative visits after a Doppler ultrasonography made by a vascular doctor in 1 month, 6 months, 12 months, 18 months and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel DAVAINE, Dr, Study Director — Pitié Salpêtrière Vascular Surgery Service
Locations (1):
- Cntre Hospitalier René Dubos, Cergy-Pontoise, France

IPD SHARING:
Plan to Share IPD: No